CLINICAL TRIAL: NCT06929767
Title: Biomarker Guided Decision-making in Acute Exacerbation of COPD: a Feasibility Study
Brief Title: Do Blood Tests Help to Decide Which Patients With Flares of Chronic Obstructive Pulmonary Disease (COPD) Need Antibiotics and Steroids?
Acronym: Bidex
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20240689-01H
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Exacerbation of COPD; AECOPD; ECOPD
Keywords: bio-maker; C reactive protein; CRP; eosinophils; exacerbation; COPD exacerbation; AECOPD; biomarker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: We are studying the use of bio-markers to aide in decision-making for the prescription of pharmacotherapy in acute exacerbations of COPD (AECOPD). The intervention arm is using bio-markers to decide whether a patient should received antibiotics and/or steroids for their AECOPD. The control arm is using standard advice from GOLD (the Global Initiative for Obstructive Lung Disease) recommendations for prescription of therapy in AECOPD.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding: The assessing physician is not blinded to group allocation, but if randomized to standard of care, the physician does not access the biomarkers (or in other words the physician writes the Rx blinded to the CRP and blood eosinophil values). The patient is blinded to group allocation and their own biomarker values but not to the specific treatment. In order to ensure the patient cannot see their own bio-markers, these results will not be released to be shared with patients in the electronic medical record. The research assistant (also the outcome assessor) will be blinded to group allocation, and biomarker values, but not to specific treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Other): If randomized to the intervention arm (biomarker-guided therapy), the physician will be provided with the biomarker-guided recommendations and will access Epic to look at the patient's biomarkers. The physician will then write a Rx for the patient keeping these recommendations in mind (but not being bound by them). Patient allergies will be taken into account when writing the Rx.
  * if blood eosinophils are >=2%, steroids are recommended
  * if blood eosinophils are < 2%, steroids are not recommended (unless the patient also has CRP < 20 with non-purulent sputum, then an abbreviated course of steroids can be considered)
  * if CRP is >= 40 mg/L,or >=20 with purulent sputum, antibiotics are recommended; if neither condition is met, antibiotics are not recommended.
  Interventions: Other: biomarker-guided decision making
- Standard of care arm (Active Comparator): If randomized to the control arm (standard of care) arm, the physician will write a prescription based on what they feel is standard of care (and will not look at the biomarker results). Patient allergies will be taken into account when writing the Rx.
  * standard of care recommendations based on most recent GOLD publication will be provided which currently include:
  * steroids in all patients with AECOPD
  * antibiotics only if there are 2 out of 3 cardinal symptoms (dyspnea, cough, sputum), and one of the symptoms has to be purulent sputum
  Interventions: Other: GOLD recommendations

INTERVENTIONS:
Other: biomarker-guided decision making — -recommendations for antibiotic and steroid Rx provided to study physician based on bio-marker (serum CRP, blood eosinophils, sputum colour) results.
  Arms: Intervention Arm
Other: GOLD recommendations — Recommendations provided to study physician for Rx of antibiotics and steroids based on current GOLD recommendations
  Arms: Standard of care arm

SUMMARY:
The goal of this clinical trial is to see if the use of two simple blood tests: C reactive protein and eosinophils, can reduce the use of steroids and antibiotics in patients with flares of chronic obstructive pulmonary disease (COPD) without reducing the chance of treatment success. Before we undertake a large trial to answer these questions, we need to do a small feasibility study to see if our study design will work. The questions we need to answer include:

How many participants will we able to include in the study over 12 months?

How many participants in the trial will take all of their medications?

Will study protocols be followed?

How much information will we be missing at the end of the study?

How many study participants will take photographs of the phlegm they are coughing up or bring in a sample of the phlegm for inspection by study doctor?

Participants will:

Come into the clinic to be assessed when they have a flare of COPD, get a chest x-ray, blood work, and a doctor visit. The doctor will provide a prescription if it is a flare of COPD.

The participant will get a call 3, 14, and 30 days later by a study researcher to ask questions about if the medications have been taken, if cough or shortness of breath remain, and if they have had to seek additional care from another doctor, clinic, or emergency room.

DETAILED DESCRIPTION:
Study design: randomized, controlled, feasibility trial

Population: Adult patients with a physician diagnosis of COPD suffering from an acute exacerbation of COPD

Intervention: Recommendations for antibiotics and/or glucocorticoids based on CRP, peripheral blood eosinophils +/- sputum colour provided to treating physician.

Comparator: Recommendations for antibiotics and/or glucocorticoids based on current standard of care recommendations in the GOLD guidelines provided to treating physician.

Recruitment/Setting: Patients with COPD will be approached in the outpatient respiratory clinic at The Ottawa Hospital during a visit to see their treating respirologist. The nurse will identify COPD patients to the treating respirologist at the beginning of the visit using coloured flags in Epic. The respirologist will ask the patient if they would like to participate in this study. If they are interested, the patient will be referred to the clinical research assistant. Alternatively, the patient can self-refer by emailing or phoning the research number on the poster. The research assistant will follow-up with the patient via telephone to discuss preferred methods of communication to discuss the trial, updates, and do the informed consent. If applicable, the research assistant will have the patient fill out a consent to communicate via email form. If the research assistant cannot reach the patient via telephone, and they initially received an email, the research assistant may respond to the email with the request that the patient sign the consent to communicate via email before any additional information is provided to the patient.

Number of Centres Participating in the feasibility study: The Ottawa Hospital only for the feasibility study.

Consent: A meeting to have the consent discussion will be coordinated by the research assistant (RA) when they first call the patient or when the patient self-refers in response to the poster. The RA will set up a video conference via MS Teams, if this is not feasible for the patient, a telephone discussion will be done. The patient will receive a copy of the consent form in advance of the meeting via either MyChart Epic, email via MS 365 Share point (download link, encrypted file), fax to their fax machine or mail (whatever they prefer). Patients will be advised that although they have verbally agreed to the trial, written consent will be obtained, and they will be asked to sign the physical consent form at the time of the in-person study visit 1.

Study Procedures

After consent, the research coordinator will provide standard education to all patients on the symptoms of AECOPD, provide them with a checklist of symptoms of AECOPD, and a phone number to call should they meet criteria for AECOPD. This phone number will be operational 8am to 11am Monday to Friday to provide a same-day in-person visit with a study respirologist (that afternoon). The patients will also be contacted via telephone or email (depending on patient preference), on the first Monday of every month to remind them of the study number to call in the event of any exacerbation. The method of communication (email or phone call) will be determined by the RA at the consent meeting. The RA will also check Epic the first Monday of each month to see if the patient was prescribed any antibiotics or prednisone outside of the trial (suggesting patient exacerbations are being missed for randomization).

If the patient experiences an AECOPD:

The patient will call the number, and the research assistant will meet the patient at the study site (at a pre-arranged location). The patient will sign the consent form. A chest x-ray and blood work (CRP, CBC with differential) will be done immediately prior to seeing the study respirologist. The study respirologist will confirm that the patient is suffering from an AECOPD (by history and physical exam) and will confirm eligibility for randomization (including ruling out fever and reviewing the chest x-ray to rule out presence of pneumonia). At this point the patient will be randomized into the study. Baseline demographics will be collected at this time including age, smoking history, last FEV1, number of exacerbations in the last year, current chronic COPD medications, use of oxygen, any positive sputum cultures within the last year. The patients will also fill out a COPD Assessment Test (CAT) score (for comparison to future values). The CAT test takes < 3 minutes to fill out.

The randomization process will consist of a computer-generated random listing of the two different treatment allocations blocked by variable blocks of two or four. Randomization will be through central allocation of a randomization schedule and will be coordinated by the Ottawa Health Research Institute.

After randomization, the treating physician will create a treatment prescription in Epic:

* If randomized to the intervention arm (biomarker-guided therapy), the physician will be provided with the biomarker-guided recommendations and will access Epic to look at the patient's biomarkers. The physician will then write a Rx for the patient keeping these recommendations in mind (but not being bound by them). Patient allergies will be taken into account when writing the Rx.
* If randomized to the control arm (standard of care) arm, the physician will write a prescription based on what they feel is standard of care (and will not look at the biomarker results). Patient allergies will be taken into account when writing the Rx.

Blinding: The assessing physician is not blinded to group allocation, but if randomized to standard of care, the physician does not access the biomarkers (or in other words the physician writes the Rx blinded to the CRP and blood eosinophil values). The patient is blinded to group allocation and their own biomarker values but not to the specific treatment. In order to ensure the patient cannot see their own bio-markers, these results will not be released to be shared with patients in the electronic medical record. The research assistant (also the outcome assessor) will be blinded to group allocation, and biomarker values, but not to specific treatment.

Assessments: Patients will be assessed at day 3, 14, and day 30 post-randomization by telephone by the clinical research assistant who is blinded to group allocation and biomarker values. At each call, requirement for additional visits for respiratory symptoms, completion of study medications, intensification or change of therapy, and the CAT will be administered. At day 3, if the patient feels worse, they will be advised to seek medical attention with their treating respirologist. The research assistant will also contact the treating respirologist to advise them of the worsening of a Bidex patient. At day 14, if the patient feels they have not improved, the research assistant will advise the patient to seek medical attention by calling their treating respirologist. The research assistant will also contact the treating respirologist to advise them of the lack of improvement of a patient enrolled in Bidex. At day 30, if the patient feels they have not improved, the research assistant will advise the patient to seek medical attention by calling their treating respirologist. The research assistant will also contact the treating respirologist to advise them of the lack of improvement of a patient enrolled in Bidex.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a known diagnosis of COPD (must have prior spirometry documenting FEV1/FVC post-bronchodilator < 0.7 or documented respirologist-diagnosis of COPD)
* Presenting with AECOPD, defined as an increase in respiratory symptoms necessitating an increase in medications
* Consent provided

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:
* new infiltrate on chest x-ray day of randomization
* temperature ≥ 38.0 ◦C taken orally day of randomization
* positive blood culture day of randomization
* co-morbid asthma or severe bronchiectasis
* acute heart failure day of randomization
* known immunosuppression including the use of chronic glucocorticoids day of randomization
* allergy/absolute contraindication to the use of oral steroids
* planned pregnancy or currently pregnant
* COVID positive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the number of patients screened, enrolled, and randomized within a 12-month period. | 12 months
  We need to know if this is a study that patients would want to do, and if this is a study that physicians would be willing to enroll or refer patients to.
  * number screened: an absolute count of patients who are contacted by the RA for initial screening and information
  * proportion enrolled: number of subjects who verbally consent divided by number of subjects screened
  * proportion randomized: number of subjects who had an exacerbation and were randomized divided by number of subjects enrolled

SECONDARY OUTCOMES:
To determine what proportion of patients had exacerbations after enrollment but prior to randomization, that were missed by the study. | 12 months
  This outcome is needed to evaluate if our method of capturing exacerbations is effective.
  -The number of times a patient was prescribed antibiotics and/or steroids between enrollment and randomization divided by number of patients enrolled.
To determine what proportion of physicians were adherent to the treatment recommendations provided. | 12 months
  To determine if physicians are willing to consider using this protocol in a study, to approximate the amount of cross-over we might get if the larger trial is not a phase 3 study
  -The number of prescriptions adherent to biomarker recommendations divided by the number of subjects randomized to the intervention arm
To determine what percentage of patients would fall into each category: What percentage had blood eosinophils > = 2% ? What percentage had CRP > = 40? What percentage had CRP < 20? What percentage had purulent sputum ? | 12 months
  To determine if we would get enough patients in all categories for a larger trial to be feasible.
  * the number of randomized subjects with blood eosinophils > =2% divided by the total number of randomized subjects
  * the number of randomized subjects with CRP > = 40 divided by total number of randomized subjects
  * the number of randomized subjects with CRP < 20 divided by the total number of randomized subjects
  * the number of randomized subjects with purulent sputum divided by the total number of randomized subjects
To determine what percentage of patients had taken a photograph of their sputum or brought sputum to be assessed in-person. | 12 months
  To determine if we would be able to reliably assess sputum purulence using this methodology in a larger trial
  -number of randomized subjects with photographs of sputum or sputum brought in container to in-person appointment divided by the total number of randomized subjects
To determine how many patients had complete data collection. | 12 months
  To determine if this protocol will provide a robust data set.
  * number of subjects with complete data set divided by number randomized.
  * complete data set includes:
  * visit 0 - CXR, blood eosinophils, CRP, CAT score
  * visit 1 - CAT score, medication adherence, questions answered re additional health care utilization
  * visit 2 - CAT score, medication adherence, questions answered re additional health care utilization
  * visit 3 - CAT score, questions answered re additional health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa PJ Luks, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramakrishnan S, Jeffers H, Langford-Wiley B, Davies J, Thulborn SJ, Mahdi M, A'Court C, Binnian I, Bright S, Cartwright S, Glover V, Law A, Fox R, Jones A, Davies C, Copping D, Russell RE, Bafadhel M. Blood eosinophil-guided oral prednisolone for COPD exacerbations in primary care in the UK (STARR2): a non-inferiority, multicentre, double-blind, placebo-controlled, randomised controlled trial. Lancet Respir Med. 2024 Jan;12(1):67-77. doi: 10.1016/S2213-2600(23)00298-9. Epub 2023 Nov 2. PMID 37924830
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Pancholi M, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Blood eosinophils to direct corticosteroid treatment of exacerbations of chronic obstructive pulmonary disease: a randomized placebo-controlled trial. Am J Respir Crit Care Med. 2012 Jul 1;186(1):48-55. doi: 10.1164/rccm.201108-1553OC. Epub 2012 Mar 23. PMID 22447964
- [Background] Zhang K, Xie K, Zhang C, Liang Y, Chen Z, Wang H. C-reactive protein testing to reduce antibiotic prescribing for acute respiratory infections in adults: a systematic review and meta-analysis. J Thorac Dis. 2022 Jan;14(1):123-134. doi: 10.21037/jtd-21-705. PMID 35242374
- [Background] Hoult G, Gillespie D, Wilkinson TMA, Thomas M, Francis NA. Biomarkers to guide the use of antibiotics for acute exacerbations of COPD (AECOPD): a systematic review and meta-analysis. BMC Pulm Med. 2022 May 13;22(1):194. doi: 10.1186/s12890-022-01958-4. PMID 35549921
- [Background] C REACTIVE PROTEIN-GUIDED ANTIBIOTIC PRESCRIBING VS STANDARD OF CARE IN EXACERBATIONS OF COPD: A SYSTEMATIC REVIEW WITH META-ANALYSIS Luks, Vanessa et al. CHEST, Volume 158, Issue 4, A1788
- [Background] Daniels JM, de Graaff CS, Vlaspolder F, Snijders D, Jansen HM, Boersma WG. Sputum colour reported by patients is not a reliable marker of the presence of bacteria in acute exacerbations of chronic obstructive pulmonary disease. Clin Microbiol Infect. 2010 Jun;16(6):583-8. doi: 10.1111/j.1469-0691.2009.02892.x. Epub 2009 Jul 20. PMID 19681947
- [Background] Brusse-Keizer MG, Grotenhuis AJ, Kerstjens HA, Telgen MC, van der Palen J, Hendrix MG, van der Valk PD. Relation of sputum colour to bacterial load in acute exacerbations of COPD. Respir Med. 2009 Apr;103(4):601-6. doi: 10.1016/j.rmed.2008.10.012. Epub 2008 Nov 22. PMID 19027281
- [Background] Stockley RA, O'Brien C, Pye A, Hill SL. Relationship of sputum color to nature and outpatient management of acute exacerbations of COPD. Chest. 2000 Jun;117(6):1638-45. doi: 10.1378/chest.117.6.1638. PMID 10858396
- [Background] Soler N, Esperatti M, Ewig S, Huerta A, Agusti C, Torres A. Sputum purulence-guided antibiotic use in hospitalised patients with exacerbations of COPD. Eur Respir J. 2012 Dec;40(6):1344-53. doi: 10.1183/09031936.00150211. Epub 2012 Apr 20. PMID 22523352
- [Background] Chen K, Pleasants KA, Pleasants RA, Beiko T, Washburn RG, Yu Z, Zhai S, Drummond MB. Procalcitonin for Antibiotic Prescription in Chronic Obstructive Pulmonary Disease Exacerbations: Systematic Review, Meta-Analysis, and Clinical Perspective. Pulm Ther. 2020 Dec;6(2):201-214. doi: 10.1007/s41030-020-00123-8. Epub 2020 Jul 16. PMID 32676981
- [Background] Li Z, Yuan X, Yu L, Wang B, Gao F, Ma J. Procalcitonin-guided antibiotic therapy in acute exacerbation of chronic obstructive pulmonary disease: An updated meta-analysis. Medicine (Baltimore). 2019 Aug;98(32):e16775. doi: 10.1097/MD.0000000000016775. PMID 31393400
- [Background] Council of the Canadian Academies, 2019. When Antibiotics Fail. Ottawa (ON). The Expert Panel on the Potential Socio-Economic Impacts of Antimicrobial Resistance in Canada, Council of Canadian Academies.
- [Background] Waljee AK, Rogers MA, Lin P, Singal AG, Stein JD, Marks RM, Ayanian JZ, Nallamothu BK. Short term use of oral corticosteroids and related harms among adults in the United States: population based cohort study. BMJ. 2017 Apr 12;357:j1415. doi: 10.1136/bmj.j1415. PMID 28404617
- [Background] Bafadhel M, Davies L, Calverley PM, Aaron SD, Brightling CE, Pavord ID. Blood eosinophil guided prednisolone therapy for exacerbations of COPD: a further analysis. Eur Respir J. 2014 Sep;44(3):789-91. doi: 10.1183/09031936.00062614. Epub 2014 Jun 12. No abstract available. PMID 24925917
- [Background] Wedzicha JA Ers Co-Chair, Miravitlles M, Hurst JR, Calverley PM, Albert RK, Anzueto A, Criner GJ, Papi A, Rabe KF, Rigau D, Sliwinski P, Tonia T, Vestbo J, Wilson KC, Krishnan JA Ats Co-Chair. Management of COPD exacerbations: a European Respiratory Society/American Thoracic Society guideline. Eur Respir J. 2017 Mar 15;49(3):1600791. doi: 10.1183/13993003.00791-2016. Print 2017 Mar. PMID 28298398
- [Background] Vollenweider DJ, Frei A, Steurer-Stey CA, Garcia-Aymerich J, Puhan MA. Antibiotics for exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2018 Oct 29;10(10):CD010257. doi: 10.1002/14651858.CD010257.pub2. PMID 30371937
- [Background] Sethi S, Evans N, Grant BJ, Murphy TF. New strains of bacteria and exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 2002 Aug 15;347(7):465-71. doi: 10.1056/NEJMoa012561. PMID 12181400
- [Background] Chen Y. Interpretation of Global Strategy for the Diagnosis, Treatment, Management and Prevention of Chronic Obstructive Pulmonary Disease 2022 Report. Vol. 25, Chinese General Practice. 2022.